CLINICAL TRIAL: NCT04222803
Title: Viral Hepatitis and Gallstone Disease Study
Acronym: VIRGAD
Status: Suspended | Type: Observational
Why Stopped: The study is currently on hold owing to the introduction of a new electronic system at some of the participating hospitals.
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Martin Lagging, MD PhD, Principal Investigator, Göteborg University
Other Study IDs: VIRGAD
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Gallstone Attack; Viral Hepatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — 9 mL serum will be sampled from each participant in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study aims to investigate possible associations between ongoing viral hepatitis (i.e. hepatitis A, B, C or E virus infection) and ultrasound or computed tomography-verified gallstone disease.

DETAILED DESCRIPTION:
Patients seeking care at emergency room at Sahlgrenska University Hospital, Gothenburg, Sweden undergoing ultrasound or computed tomography for suspected gallstone disease, will be asked if they wish to participate in the study. If they agree, a serum sample will be draw for analysis of anti-HAV IgM, HBsAg, anti-HCV, HCV Core antigen and HEV RNA. The proportion of patients with vs. without ultrasound or computed tomography-verified gallstone disease will be evaluated regarding possible ongoing viral hepatitis (i.e. hepatitis A, B, C or E virus infection).

ELIGIBILITY:
Inclusion Criteria:

* Acute abdominal pain entailing an abdominal ultrasound or computed tomography for suspected gallstone disease at the emergency room at Sahlgrenska University Hospital, Gothenburg
* Written informed consent
* Ability to obtain 9 mL serum for analysis of anti-HAV IgM, HBsAg, anti-HCV, HCV Core antigen and HEV RNA

Exclusion Criteria:

* Not willing to give written informed consent
* Age below 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without ultrasound or computed tomography-verified gallstone disease will be compared for biomarkers of ongoing viral hepatitis (i.e. anti-HAV IgM, HBsAg, HCV Core antigen and HEV RNA).
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2027-10-09 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between ongoing viral hepatitis (i.e. hepatitis A, B, C or E virus infection) and ultrasound or computed tomography-verified gallstone disease | 1 day
  The proportion of patient with verified gallstone disease having detectable anti-HAV IgM, HBsAg, HCV Core antigen or HEV RNA will be compared with the proportion among patients without verified gallstone disease.
Association between ongoing hepatitis A virus infection and ultrasound or computed tomography-verified gallstone disease | 1 day
  The proportion of patient with verified gallstone disease having detectable anti-HAV IgM will be compared with the proportion among patients without verified gallstone disease.
Association between ongoing hepatitis B virus infection and ultrasound or computed tomography-verified gallstone disease | 1 day
  The proportion of patient with verified gallstone disease having detectable HBsAg will be compared with the proportion among patients without verified gallstone disease.
Association between ongoing hepatitis C virus infection and ultrasound or computed tomography-verified gallstone disease | 1 day
  The proportion of patient with verified gallstone disease having detectable HCV Core antigen will be compared with the proportion among patients without verified gallstone disease.
Association between ongoing hepatitis E virus infection and ultrasound or computed tomography-verified gallstone disease | 1 day
  The proportion of patient with verified gallstone disease having detectable HEV RNA will be compared with the proportion among patients without verified gallstone disease.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Martin, MD PhD, Principal Investigator — Göteborg University
Locations (1):
- Södra Älvsborgs Sjukhus, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No